CLINICAL TRIAL: NCT00902031
Title: Randomized, Double-Blind, Placebo-Controlled Trial of Oral Docusate for Preventing/Treating Constipation in Palliative Care Patients.
Brief Title: Effectiveness of Docusate in Preventing/Treating Constipation in Palliative Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: College of Family Physicians of Canada (Other); Covenant Health, Canada (Other); Capital Care (Unknown)
Responsible Party: Dr. Richard Spooner, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: G599001036; G517000014
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Constipation; Palliative Care
Keywords: Docusate; Constipation; Colace; Palliative Care; Sennoside; Senokot; Terminally Ill; Stool; Randomized Trial
MeSH Terms: conditions — Constipation | interventions — Dioctyl Sulfosuccinic Acid; Sennosides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docusate + Sennoside (Experimental)
  Interventions: Drug: Docusate Sodium, Sennoside
- Sennoside + Placebo (Placebo Comparator)
  Interventions: Drug: Sennoside + Placebo

INTERVENTIONS:
Drug: Docusate Sodium, Sennoside — Docusate sodium: given in capsule form (100 mg/capsule), at a dosage of 200 mg, taken twice daily for 10 days.
  Sennoside: will be given in tablet form (8.6 mg), 1-3 tablets taken 1-3 times daily for 10 days.
  Other Names: Colace; Senokot
  Arms: Docusate + Sennoside
Drug: Sennoside + Placebo — Sennoside: will be given in tablet form (8.6 mg), 1-3 tablets taken 1-3 times daily for 10 days.
  Placebo: will be taken in capsule form, similar in size, shape, and color to docusate, taken twice daily for 10 days
  Other Names: Senokot
  Arms: Sennoside + Placebo

SUMMARY:
The purpose of this study is to determine if docusate is effective in the treatment of constipation in palliative care patients.

DETAILED DESCRIPTION:
Palliative patients frequently experience constipation due to multiple factors - structural abnormalities, medications, metabolic disturbances, neurological disorders, and other general conditions. Docusate is a stool softener that has been widely used, in combination with other stimulating laxatives, to prevent and treat constipation in palliative care patients. In the past decade there has been controversy about its effectiveness in these populations, but no controlled trials have been conducted on the use of docusate in palliative patients. The purpose of this study is to assess the effectiveness of docusate in preventing and treating constipation in palliative care patients. The study design is a randomized, double-blind, placebo-controlled trial to compare the current standard treatment (docusate in combination with a laxative, sennoside) to that of a sennoside laxative alone. A total of 70 patients (35 in each group) will be recruited from the Palliative Care Unit at St. Joseph's Auxiliary Care Hospital, the Mel Miller Hospice at the Edmonton General Continuing Care Hospital, and CapitalCare Norwood in Edmonton, Alberta, Canada. Patients must be ≥ 18 years of age, able to take oral medication, without difficulty swallowing, have a palliative performance ≥ 20%, and do not have a stoma. The duration of treatment will be for 10 days. The main outcome measures will include bowel frequency, stool consistency, other interventions (suppositories, enemas), difficulty defecating, and sense of inability to evacuate completely. This study will provide insight into the effectiveness of docusate in preventing and treating constipation in palliative patients who are cared for by family physicians and specialized palliative care providers. If docusate is found to have no added benefit,it has the potential to enhance the quality of life for palliative care patients by reducing the number of medications taken and reducing the palliative care team's (e.g. nursing) workload and cost.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years of age
* new admissions
* able to take oral medications
* patient and/or personal directive agent (proxy) provides written consent
* does not have a stoma
* no difficulty swallowing
* no previous intolerance/contraindications to docusate
* palliative performance greater than or equal to 20%

Exclusion Criteria:

* less than 18 years of age
* failing to provide consent
* unable to take oral medication/difficulty swallowing
* previous intolerance/contraindications to docusate (Colace)
* patients who have a stoma
* palliative performance status < 20%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2006-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Stool Frequency | 10 days
Stool Consistency | 10 day
Difficulty Defecating | 10 day
Symptoms Related to Constipation (pain, nausea, appetite loss, abdominal discomfort, shortness of breath) | 10 day
Type of Additional Bowel Care Interventions which may be Required | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Spooner, MD, Principal Investigator — University of Alberta; Yoko Tarumi, MD, Principal Investigator — University of Alberta/Regional Palliatvie Care Program (Capital Health); Olga Szafran, MSc., Study Director — University of Alberta
Locations (3):
- Canada (3):
  - CapitalCare Norwood, Edmonton, Alberta
  - Mel Miller Hospice at Edmonton General Continuing Care Hospital, Edmonton, Alberta
  - St. Joseph's Auxiliary Care Hospital, Edmonton, Alberta

REFERENCES:
- [Background] CASS LJ, FREDERIK WS. Doxinate in the treatment of constipation. Am J Gastroenterol. 1956 Dec;26(6):691-8. No abstract available. PMID 13372512
- [Background] Castle SC, Cantrell M, Israel DS, Samuelson MJ. Constipation prevention: empiric use of stool softeners questioned. Geriatrics. 1991 Nov;46(11):84-6. No abstract available. PMID 1718823
- [Background] Fain AM, Susat R, Herring M, Dorton K. Treatment of constipation in geriatric and chronically ill patients: a comparison. South Med J. 1978 Jun;71(6):677-80. doi: 10.1097/00007611-197806000-00022. PMID 78527
- [Background] Goodman J, Pang J, Bessman AN. Dioctyl sodium sulfosuccinate- an ineffective prophylactic laxative. J Chronic Dis. 1976 Jan;29(1):59-63. doi: 10.1016/0021-9681(76)90068-0. No abstract available. PMID 1254685
- [Background] Hurdon V, Viola R, Schroder C. How useful is docusate in patients at risk for constipation? A systematic review of the evidence in the chronically ill. J Pain Symptom Manage. 2000 Feb;19(2):130-6. doi: 10.1016/s0885-3924(99)00157-8. PMID 10699540